CLINICAL TRIAL: NCT04386460
Title: Covid-19 and Prevention of Malnutrition After Confinement by Dentists: Prospective Study Among 100 Adults Received in Dental Consultation at Nice University Hospital and Sent to Their Physician for Assessment and Nutritional Care
Brief Title: Covid-19 and Prevention of Malnutrition After Confinement by Dentists
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Other Study IDs: 20odontocovid-02
Record Dates: First submitted 2020-05-12; First posted 2020-05-13 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2020-05

CONDITIONS: Nutrition Poor; Infection Viral; Oral Disease
MeSH Terms: conditions — Malnutrition; Virus Diseases; Mouth Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Background. The Covid-19 pandemic reached France in January 2020 and the French government decreed the confinement of the population for eight weeks, from March 17 to May 10, 2020. Dental surgeries were closed and only dental emergency services were provided. Dental surgeries reopened on May 11th, with a limited focus on urgent care, by applying new occupational hygiene standards to limit the circulation of SARS-Cov-2 coronavirus. Hypothesis. From May 11th, chronic patients and elderly patients who come to the hospital for dental consultations will have two risks of malnutrition:

DETAILED DESCRIPTION:
Background. The Covid-19 pandemic reached France in January 2020 and the French government decreed the confinement of the population for eight weeks, from March 17 to May 10, 2020. Dental surgeries were closed and only dental emergency services were provided. Dental surgeries reopened on May 11th, with a limited focus on urgent care, by applying new occupational hygiene standards to limit the circulation of SARS-Cov-2 coronavirus. Hypothesis. From May 11th, chronic patients and elderly patients who come to the hospital for dental consultations will have two risks of malnutrition:

1) because of confinement (loneliness, anorexia, difficulty shopping) and 2) because of the untreated dental problem (oral pain or untreated edentulism). Main objective. To investigate whether dentists' recommendation to consult a physician is efficient to prevent or to treat malnutrition. Secondary objective. Conduct a medico-economic study to assess the health savings generated by the prevention of malnutrition by dentists. Type of study and population studied. Prospective cohort study including 100 adults received in hospital dental consultation, malnourished or at risk of malnutrition. Inclusion criteria. All subjects answering "yes" to one of these two questions: 1) "Do you eat less?" and/or 2) "Have you lost weight?" Exclusion criteria. None. Study design and evaluation criteria. At baseline, for all subjects included, the dentist will check the weight (kg, weighed), the usual weight (kg, question), height (m, question or from ID card), masticatory ability (score 0%-100%) and oral pain (score 0-10). Then the dentist will give the patient a note advising him to consult his doctor for assessment and management of malnutrition. The dentist will call the patient 1 month (M1) and 3 months (M3) after baseline, to ask him for his weight (kg), if he consulted his doctor (yes/no) and received nutritional supplements (if yes, what prescription). Main evaluation criterion. Body Mass Index (BMI kg/m²) evolution from baseline to M1 and M3. Secondary evaluation criteria. Weight changes during confinement, medical consultation, prescription of nutritional supplements and observance. Individual duration of the study. Three months. Total duration of the study. One year. Expected fallout. To improve the nutritional status of malnourished participants, following confinement. To anticipate malnutrition in exposed populations in the case of a second viral pandemic and confinement. Educate dentists on the importance of screening and managing malnutrition in at-risk patients.

ELIGIBILITY:
Inclusion Criteria:

* All subjects answering "yes" to one of these two questions: 1) "Do you eat less?" and/or 2) "Have you lost weight?"

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patient in University hospital dental clinic
Sampling Method: Non-Probability Sample
Enrollment: 17 (Actual)
Dates: Start 2020-05-11 (Actual); Primary Completion 2020-06-05 (Actual); Study Completion 2021-05-11 (Actual)

PRIMARY OUTCOMES:
Body Mass Index | 1 Month
  Body Mass Index evolution from baseline
Body Mass Index | 3 Months
  Body Mass Index evolution from baseline

SECONDARY OUTCOMES:
Weight changes during confinement | 8 weeks
  Usual weight at baseline vs weight before confinement (gk)
prescription of nutritional supplements and observance | 3 months
  number and type of nutritional supplements from baseline

CONTACTS AND LOCATIONS:
Locations (1):
- University Nice Hospital, Nice, France